CLINICAL TRIAL: NCT06411730
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered BMS-986368 in Healthy Participants, Healthy Elderly Participants, and Healthy Participants of Japanese Ethnicity
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of Orally Administered BMS-986368 in Healthy Participants, Healthy Elderly Participants, and Healthy Participants of Japanese Ethnicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IM045-1009
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Pharmacodynamics; BMS-986368; CC-97489; Healthy Volunteers; Elderly Volunteers; Japanese Volunteers; Multiple Ascending Dose; Healthy Participants; Elderly Participants; Japanese Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1A (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 1B (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 1C (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 2A (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 2B (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 2C (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 2D (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 3A (Experimental)
  Interventions: Drug: BMS-986368
- Cohort 3B (Experimental)
  Interventions: Drug: BMS-986368

INTERVENTIONS:
Drug: BMS-986368 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of orally administered BMS-986368 in healthy participants, healthy elderly participants, and healthy participants of japanese ethnicity.

ELIGIBILITY:
Inclusion Criteria

* Participants must be healthy male or non-pregnant and non-nursing female individuals.
* For Part 2 only, participants must be of Japanese ethnicity (both biological parents are ethnically Japanese).
* Participants must have a body mass index (BMI) of 18.0 kg/m2 to 33.0 kg/m2, inclusive.
* Participants must have normal renal function at screening.

Exclusion Criteria

* Participants must not have a personal or first-degree family (individual's parents, siblings, and children) history of clinically significant psychiatric disorder, including, but not limited to, schizophrenia, psychosis, bipolar disorder, panic disorder, generalized anxiety disorder, and obsessive-compulsive disorder.
* Participants must not have any significant acute or chronic neurological illness (eg, history of intracranial or intraspinal hemorrhage, CNS lesions, recent bacterial or fungal meningitis, etc) as determined by the investigator.
* Participants must not have a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary (GU) abnormalities/diseases including but not limited to peptic ulcer disease, or significant GI bleeding, pancreatitis, hypokalemia.
* Participants must not have had a SARS-CoV-2 infection within 2 weeks prior to screening.
* Participants must not have a history of any significant drug allergy or hypersensitivity (such as anaphylaxis or hepatotoxicity).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 44 days
Number of participants with serious adverse events (SAEs) | Up to 44 days
Number of participants with vital sign (VS) abnormalities | Up to 21 days
Number of participants with physical examination abnormalities | Up to 21 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 21 days
Number of participants with clinical laboratory asssement abnormalities | Up to 21 days
Number of participants with treatment-emergent suicidal ideation and behavior through assessment of Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 21 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Up to 16 days
Maximum observed plasma concentration (Cmax) | Up to 16 days
Time of maximum observed plasma concentration (Tmax) | Up to 16 days
Absolute levels of monoacylglycerol lipase (MGLL) enzymatic activities in peripheral blood mononuclear cells (PBMCs) | Up to 21 days
Percent change from baseline for monoacylglycerol lipase (MGLL) enzymatic activities in peripheral blood mononuclear cells (PBMCs) | Up to 21 days
Plasma concentrations of anandamide (AEA) | Up to 21 days
Percent change from baseline of anandamide (AEA) | Up to 21 days
Whole blood concentrations of 2-arachidonoylglycerol (2-AG) | Up to 21 days
Percent change from baseline of 2-arachidonoylglycerol (2-AG) | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com